CLINICAL TRIAL: NCT05698732
Title: Coroflex® ISAR NEO Coronary Stent System Post-Market Clinical Follow-up Study
Brief Title: Coroflex® ISAR NEO PMCF Study
Acronym: rEPIC07
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: Coroflex® ISAR NEO PMCF Study
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Disease (CAD) and high risk of bleeding
  Interventions: Device: Coroflex® ISAR NEO coronary stent system
- Coronary Artery Disease (CAD)
  Interventions: Device: Coroflex® ISAR NEO coronary stent system

INTERVENTIONS:
Device: Coroflex® ISAR NEO coronary stent system — Patients in whom treatment with Coroflex® ISAR NEO coronary stent system has been attempted

SUMMARY:
International, Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Coroflex® ISAR NEO coronary stent system to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Coroflex® ISAR NEO coronary stent system sirolimus eluting stent.

DETAILED DESCRIPTION:
The objective of this international, multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the Coroflex® ISAR NEO coronary stent system Sirolimus Eluting Stent in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

Coroflex® ISAR NEO is intended to be used for

* Patients must be at least 18 years of age AND
* The patient must fulfill the standard recommendations for Percutaneous Coronary Intervention (PCI) based on the last European Society of Cardiology (ESC) recommendations within his/ her regular treatment or that the use of the product has already been decided within the regular planning of the patient's treatment AND
* Patients with Novo lesion length 2-4 mm AND
* Informed consent signed

Exclusion Criteria:

* Patients with express refusal by the patient to participate in the study.
* Patients pregnant women and lactating women.
* Patients with acute coronary syndrome (ACS) in a situation of cardiogenic shock (Killip 4).
* Patients in whom anti-platelet and/or anti-coagulation therapy is contraindicated
* Patients with lesions, that possibly can not be treated successfully with Percutaneous transluminal Coronary Angioplasty (PTCA) or stent implantation
* Patients with known sensitivity to Sirolimus, the carrier Probucol, the procedural co-medication or the alloying component of the stent
* Patients with known sensitivity to contrast agents who cannot be premedicated.
* Patients with contraindications or hypersensitivity to sirolimus
* Patients with a life expectancy of less than 2 years
* Patients included in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Coroflex® ISAR NEO coronary stent system according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, stent thrombosis (Academic Research Consortium definitive/ probable), and new Target Lesion Revascularization (TLR)
Efficacy Endpoint. Freedom fromTarget Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Freedom from Accidental dislodgement of the stent | During percutaneous coronary intervention (PCI)
  Freedom from Accidental dislodgement of the stent
Freedom from Balloon rupture | During PCI
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI
  Freedom from Hypotube rupture
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (18):
- France (6):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre Hospitalier Ajaccio, Ajaccio
  - University Hospital Center of Caen, Caen
  - Hôpital Albert Schweitzer, Colmar
  - Hospitalario Universitario (CHU) de Lille, Lille
  - APHP -Hôpital Lariboisière, Paris
- Spain (12):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario San Pedro de Alcantara, Cáceres
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Leon, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Urban P, Mehran R, Colleran R, Angiolillo DJ, Byrne RA, Capodanno D, Cuisset T, Cutlip D, Eerdmans P, Eikelboom J, Farb A, Gibson CM, Gregson J, Haude M, James SK, Kim HS, Kimura T, Konishi A, Laschinger J, Leon MB, Magee PFA, Mitsutake Y, Mylotte D, Pocock S, Price MJ, Rao SV, Spitzer E, Stockbridge N, Valgimigli M, Varenne O, Windhoevel U, Yeh RW, Krucoff MW, Morice MC. Defining high bleeding risk in patients undergoing percutaneous coronary intervention: a consensus document from the Academic Research Consortium for High Bleeding Risk. Eur Heart J. 2019 Aug 14;40(31):2632-2653. doi: 10.1093/eurheartj/ehz372. PMID 31116395
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Ruiz-Nodar JM, Ferreiro JL. Tratamiento antitrómbotico tras revascularización percutánea en pacientes con indicación crónica de anticoagulación oral. REC Interv Cardiol. 2019;1(1):41-50.